CLINICAL TRIAL: NCT00132522
Title: A Study to Find the Highest Dose of Biological Study Drug (EMD 273066) That Can Be Given Safely to Patients With Recurrent EpCAM Positive Ovarian, Prostate, Colorectal or Non-Small Cell Lung Cancers When First Given a Low Dose of Cyclophosphamide
Brief Title: EMD 273066 in Patients With Recurrent EpCAM Positive Ovarian, Prostate, Colorectal or Non-small Cell Lung Cancers When First Given Cyclophosphamide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62206-015
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Ovarian Cancer; Colorectal Cancer; Carcinoma, Non-small-cell Lung; Prostate Cancer
Keywords: EpCAM; monoclonal-antibody; targeted therapy; colorectal; prostate; non-small cell lung cancer; ovarian; solid tumor
MeSH Terms: conditions — Ovarian Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms | interventions — tucotuzumab celmoleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: EMD 273066

INTERVENTIONS:
Drug: EMD 273066 — dose-escalating study and subjects enrolled in the study may receive a maximum of 6 cycles of the assigned regimen over 18 weeks. Each cycle will be 3 weeks (21 days) with cyclophosphamide on Day 1 and EMD 273066 on Days 2 to 4, followed by 17 days with no experimental pharmaceutical product.
  Each cycle, cyclophosphamide at 300 mg/m2 given per institutional guidelines 1 day (22-28 hours) prior to 3 consecutive days of EMD 273066 as a 4-hour IV infusion at 1 of 6 planned dose levels of 0.5, 1, 2, 3, 4, or 6 mg/m2.

SUMMARY:
This study is looking at the safety and tolerability of the experimental biological drug EMD 273066 when given with low dose cyclophosphamide to patients with recurring EpCAM positive ovarian, prostate, colorectal or non-small cell lung cancers. EMD 273066 is an experimental biological drug that may increase the immune response to certain cancers. Patients will be enrolled in groups of 3, with each successive group receiving a higher dose if the prior group adequately tolerates the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent non-small cell lung, colorectal, ovarian or prostate cancer
* No more than two lines of prior chemotherapy
* Positive EpCAM expression
* Karnofsky Performance Status > 70%
* Adequate laboratory results
* Normal cardiac stress test

Exclusion Criteria:

* Evidence of brain metastases
* Pregnant or lactating females
* Significant infection
* Prior receipt of EMD 273066
* Unable to interrupt anti-hypertensive medications 2 days prior to and through each cycle of study medication administration
* Uncontrolled hypertension
* Previous diagnosis of Addison's disease
* Previous diagnosis of an autoimmune disease
* Organ transplant
* Insulin-dependent diabetes
* History of acute pancreatitis
* Congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-05; Primary Completion 2008-06 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
efficacy | various timepoints
safety | various timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Joseph O'Connor, MD, Principal Investigator — University of Wisconsin, Madison
Locations (5):
- United States (4):
  - City of Hope, Durate, California
  - Dartmouth Medical School, Pharmacology & Toxicology Dept. of Medicine, Lebanon, New Hampshire
  - Fox Chase Cancer Oncology Department of Medical Oncology, Philadelphia, Pennsylvania
  - University of Wisconsin Division of Gynecologic Oncology, Madison, Wisconsin
- Centre pluridisciplinaire d'Oncologie, Lausanne, Rue Du Bugnon, Switzerland

REFERENCES:
- [Derived] Connor JP, Cristea MC, Lewis NL, Lewis LD, Komarnitsky PB, Mattiacci MR, Felder M, Stewart S, Harter J, Henslee-Downey J, Kramer D, Neugebauer R, Stupp R. A phase 1b study of humanized KS-interleukin-2 (huKS-IL2) immunocytokine with cyclophosphamide in patients with EpCAM-positive advanced solid tumors. BMC Cancer. 2013 Jan 15;13:20. doi: 10.1186/1471-2407-13-20. PMID 23320927